CLINICAL TRIAL: NCT00021255
Title: Multicenter Phase III Randomized Trial Comparing Doxorubicin and Cyclophosphamide Followed By Docetaxel (AC-T) With Doxorubicin and Cyclophosphamide Followed By Docetaxel and Trastuzumab (Herceptin)(AC-TH) and With Docetaxel, Carboplatin and Trastuzumab (TCH) In The Adjuvant Treatment Of Node Positive and High Risk Node Negative Patients With Operable Breast Cancer Containing The HER2 Alteration
Brief Title: Combination Chemotherapy With or Without Trastuzumab in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Cancer International Research Group (CIRG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAX_GMA_302; BCIRG 006; NCT00768092 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-09

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Docetaxel; Trastuzumab; Carboplatin

ARMS (3):
- Doxorubicin+Cyclophosphamide (AC) followed by Docetaxel (AC→T) (Experimental): Doxorubicin 60 mg/m² intravenous (IV) bolus injection in combination with cyclophosphamide 600 mg/m² IV bolus injection on Day 1 of every 3 weeks for 4 cycles followed by docetaxel 100 mg/m² IV infusion every 3 weeks for another 4 cycles.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel
- AC followed by Docetaxel + Herceptin (AC→TH) (Experimental): Doxorubicin 60 mg/m² IV bolus injection in combination with cyclophosphamide 600 mg/m² IV bolus Injection on Day 1 of every 3 weeks for 4 cycles. Herceptin 4 mg/kg IV infusion on Day 1 of Cycle 5, followed by Herceptin 2 mg/kg by IV infusion weekly starting from Day 8; and docetaxel 100 mg/m² IV infusion on Day 2 of Cycle 5, then on Day 1 of every 3 weeks for all subsequent cycles ( total 4 cycles). After completion of the last cycle of chemotherapy, Herceptin 6 mg/kg IV infusion was administered every 3 weeks until 1 year from date of initial Herceptin dose.
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Herceptin
- Docetaxel + Carboplatin + Herceptin (TCH) (Experimental): Herceptin 4 mg/kg IV infusion on Day 1 of Cycle 1 only, followed by Herceptin 2 mg/kg IV infusion weekly starting from Day 8 until three weeks after the last cycle of chemotherapy. Docetaxel 75 mg/ m² IV infusion on Day 2 of Cycle 1, then on Day 1 of all subsequent cycles followed by carboplatin IV infusion at target AUC = 6 mg/mL/min repeated every 3 weeks for a total of 6 cycles. After completion of the last cycle of chemotherapy, Herceptin 6 mg/kg by IV infusion was administered every 3 weeks until 1 year from date of initial Herceptin dose.
  Interventions: Drug: Docetaxel; Drug: Herceptin; Drug: Carboplatin

INTERVENTIONS:
Drug: Doxorubicin
  Arms: AC followed by Docetaxel + Herceptin (AC→TH); Doxorubicin+Cyclophosphamide (AC) followed by Docetaxel (AC→T)
Drug: Cyclophosphamide
  Arms: AC followed by Docetaxel + Herceptin (AC→TH); Doxorubicin+Cyclophosphamide (AC) followed by Docetaxel (AC→T)
Drug: Docetaxel
  Other Names: Taxotere
Drug: Herceptin
  Other Names: Trastuzumab
  Arms: AC followed by Docetaxel + Herceptin (AC→TH); Docetaxel + Carboplatin + Herceptin (TCH)
Drug: Carboplatin
  Arms: Docetaxel + Carboplatin + Herceptin (TCH)

SUMMARY:
Primary objective:

* Compare disease-free survival in women with human epidermal growth factor receptor 2 (HER2)-neu-expressing node-positive or high-risk node-negative operable breast cancer treated with adjuvant doxorubicin, cyclophosphamide, and docetaxel with or without trastuzumab (Herceptin) vs trastuzumab, docetaxel, and carboplatin.

Secondary objective:

* Compare overall survival of participants treated with these regimens.
* Compare the toxic effects (including cardiac) of these regimens in these participants.
* Compare quality of life of participants treated with these regimens.
* Compare pathologic and molecular markers for predicting efficacy of these regimens in these participants.
* For substudy: Compare peripheral levels of shed HER2-neu extracellular domain with fluorescence in situ hybridization in predicting outcome in participants treated with these regimens.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the participants for treatment and follow-up.
* Accessible for treatment and follow-up at participating centers.
* Histologically proven breast cancer with an interval between definitive surgery that included axillary lymph node involvement assessment and registration of less than or equal to 60 days. A central pathology review might be performed post randomization for confirmation of diagnosis and molecular studies. The same block used for HER2neu determination prior to randomization might be used for the central pathology review.
* Definitive surgical treatment must be either mastectomy with axillary lymph node involvement assessment, or breast conserving surgery with axillary lymph node involvement assessment for operable breast cancer (T1-3, Clinical N0-1, M0). Margins of resected specimen from definitive surgery must be histologically free of invasive adenocarcinoma and/or ductal carcinoma in situ (DCIS).
* Participants must be either lymph node positive or high risk node negative. Lymph node positive participants were to be defined as participants having invasive adenocarcinoma with at least one axillary lymph node (pN1) showing evidence of tumor among a minimum of six resected lymph nodes. High risk lymph node negative participants were to be defined as participants having invasive adenocarcinoma with either 0 (pNo) among a minimum of 6 resected lymph nodes or negative sentinel node biopsy (pNo) and at least one of the following factors: tumor size > 2 cm, estrogen receptor (ER) and/or progesteron receptor (PR) status was negative, histologic and/or nuclear grade 2-3, or age < 35 years.
* Tumor must show the presence of the HER2neu gene amplification by Fluorescence In-Situ Hybridization (FISH analysis) by a designated central laboratory.
* Estrogen and/or progesterone receptor analysis performed on the primary tumor prior to randomization. Results must be known at the time of randomization.
* Karnofsky Performance status index ≥ 80%.
* Normal cardiac function must be confirmed by left ventricular ejection fraction (LVEF) (multiple-gated acquisition [MUGA] scan) and electrocardiogram (ECG) within 3 months prior to registration. The result of the MUGA must be equal to or above the lower limit of normal for the institution.
* Laboratory requirements: (within 14 days prior to registration)

  a) Hematology: i) Neutrophils ≥ 2.0 109/L ii) Platelets ≥ 100 109/L iii) Hemoglobin ≥ 10 g/Dl

  b) Hepatic function: i) Total bilirubin ≤ 1 UNL ii) Aspartate aminotransferase (ASAT) (Serum glutamic oxaloacetic transaminase [SGOT]) and alanine amino transferase (ALAT) (Serum glutamic-pyruvic transaminase [SGPT]) ≤ 2.5 UNL iii) Alkaline phosphatase ≤ 5 UNL iv) Participants with ASAT and/or ALAT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL are not eligible for the study.

  c) Renal function: i) Creatinine ≤ 175 µmol/L (2 mg/dL) ii) If creatinine was 140 - 175 μmol/L, the calculated creatinine clearance should be ≥ 60 mL/min.
* Complete staging work-up within 3 months prior to registration. All participants had bilateral mammography, chest X-ray (posterioanterior [PA] and lateral) and/or computerized tomography (CT) and/or magnetic resonance imaging (MRI), abdominal ultrasound and/or CT scan and/or MRI, and bone scan. In cases of positive bone scans, bone X-ray evaluation was mandatory to rule out the possibility of metastatic bone scan positivity. Other tests may be performed as clinically indicated.
* Negative pregnancy test (urine or serum) within 7 days prior to registration for all women of childbearing potential.
* An audiology assessment with normal results was to be performed within 4 weeks of registration. This was only for those centers who had selected cisplatin as their platinum salt of choice for the BCIRG 006 study.

Exclusion criteria:

* Prior systemic anticancer therapy for breast cancer (immunotherapy, hormonotherapy, chemotherapy).
* Prior anthracycline therapy, taxoids (paclitaxel, docetaxel) or platinum salts for any malignancy.
* Prior radiation therapy for breast cancer.
* Bilateral invasive breast cancer.
* Pregnant, or lactating participants. Participants of childbearing potential must implement adequate non-hormonal contraceptive measures during study treatment (chemotherapy and tamoxifen therapy) and must had negative urine or serum pregnancy test within 7 days prior to registration.
* Any T4 or N2 or known N3 or M1 breast cancer.
* Pre-existing motor or sensory neurotoxicity of a severity ≥ grade 2 by National Cancer Institute (NCI) criteria.
* Cardiac disease that would preclude the use of doxorubicin, docetaxel and Herceptin:

  1. any documented myocardial infarction
  2. angina pectoris that required the use of antianginal medication
  3. any history of documented congestive heart failure
  4. Grade 3 or Grade 4 cardiac arrhythmia (NCI Common Terminology Criteria [CTC], version 2.0)
  5. clinically significant valvular heart disease
  6. participants with cardiomegaly on chest x-ray or ventricular hypertrophy on ECG, unless they demonstrate by MUGA scan within the past 3 months that the LVEF was ≥ the lower limit of normal for the radiology facility;
  7. participants with poorly controlled hypertension i.e. diastolic greater than 100 mm/Hg. (Participants who were well controlled on medication were eligible for entry)
  8. participants who currently received medications (digitalis, beta-blockers, calcium channel-blockers, etc) that altered cardiac conduction, if these medications were administered for cardiac arrhythmia, angina or congestive heart failure. If these medications were administered for other reasons (ie hypertension), the participant was eligible.
* Other serious illness or medical condition:

  1. history of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent
  2. active uncontrolled infection
  3. active peptic ulcer, unstable diabetes mellitus
  4. impaired hearing (only for those participants treated at centers who had selected cisplatin as their platinum salt of choice)
* Past or current history of neoplasm other than breast carcinoma, except for:

  1. curatively treated non-melanoma skin cancer
  2. in situ carcinoma of the cervix
  3. other cancer curatively treated and with no evidence of disease for at least 10 years
  4. ipsilateral DCIS of the breast
  5. lobular carcinoma in-situ (LCIS) of the breast
* Current therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators (SERMs), either for osteoporosis or prevention. Participants must had discontinued these agents prior to randomization.
* Chronic treatment with corticosteroids unless initiated > 6 months prior to study entry and at low dose (≤ 20 mg methylprednisolone or equivalent).
* Concurrent treatment with ovarian hormonal replacement therapy. Prior treatment must be stopped prior to randomization.
* Definite contraindications for the use of corticosteroids.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
* Concurrent treatment with any other anti-cancer therapy.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3222 (Actual)
Dates: Start 2001-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AUSSEL Jean Philippe, Study Director — Sanofi
Locations (42):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Sarajevo, Bosnia and Herzegovina
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Vazrjdane Region, Bulgaria
- Sanofi-Aventis Administrative Office, Québec, Canada
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Frankfurt, Germany
- Sanofi-Aventis Administrative Office, Kallithea, Greece
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Dublin, Ireland
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Beirut, Lebanon
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico
- Sanofi-Aventis Administrative Office, Macquarie Park, New Zealand
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Ljubljana, Slovenia
- Sanofi-Aventis Administrative Office, Gauteng, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom
- Sanofi-Aventis Administrative Office, Montevideo, Uruguay
- Sanofi-Aventis Administrative Office, Caracas, Venezuela

REFERENCES:
- [Background] Slamon D, Eiermann W, Robert N, Pienkowski T, Martin M, Press M, Mackey J, Glaspy J, Chan A, Pawlicki M, Pinter T, Valero V, Liu MC, Sauter G, von Minckwitz G, Visco F, Bee V, Buyse M, Bendahmane B, Tabah-Fisch I, Lindsay MA, Riva A, Crown J; Breast Cancer International Research Group. Adjuvant trastuzumab in HER2-positive breast cancer. N Engl J Med. 2011 Oct 6;365(14):1273-83. doi: 10.1056/NEJMoa0910383. PMID 21991949
- [Background] Au HJ, Eiermann W, Robert NJ, Pienkowski T, Crown J, Martin M, Pawlicki M, Chan A, Mackey J, Glaspy J, Pinter T, Liu MC, Fornander T, Sehdev S, Ferrero JM, Bee V, Santana MJ, Miller DP, Lalla D, Slamon DJ; Translational Research in Oncology BCIRG 006 Trial Investigators. Health-related quality of life with adjuvant docetaxel- and trastuzumab-based regimens in patients with node-positive and high-risk node-negative, HER2-positive early breast cancer: results from the BCIRG 006 Study. Oncologist. 2013;18(7):812-8. doi: 10.1634/theoncologist.2013-0091. Epub 2013 Jun 28. PMID 23814044
- [Background] Perez EA, Press MF, Dueck AC, Jenkins RB, Kim C, Chen B, Villalobos I, Paik S, Buyse M, Wiktor AE, Meyer R, Finnigan M, Zujewski J, Shing M, Stern HM, Lingle WL, Reinholz MM, Slamon DJ. Immunohistochemistry and fluorescence in situ hybridization assessment of HER2 in clinical trials of adjuvant therapy for breast cancer (NCCTG N9831, BCIRG 006, and BCIRG 005). Breast Cancer Res Treat. 2013 Feb;138(1):99-108. doi: 10.1007/s10549-013-2444-y. Epub 2013 Feb 19. PMID 23420271
- [Background] Press MF, Sauter G, Buyse M, Bernstein L, Guzman R, Santiago A, Villalobos IE, Eiermann W, Pienkowski T, Martin M, Robert N, Crown J, Bee V, Taupin H, Flom KJ, Tabah-Fisch I, Pauletti G, Lindsay MA, Riva A, Slamon DJ. Alteration of topoisomerase II-alpha gene in human breast cancer: association with responsiveness to anthracycline-based chemotherapy. J Clin Oncol. 2011 Mar 1;29(7):859-67. doi: 10.1200/JCO.2009.27.5644. Epub 2010 Dec 28. PMID 21189395
- [Background] Stern HM, Gardner H, Burzykowski T, Elatre W, O'Brien C, Lackner MR, Pestano GA, Santiago A, Villalobos I, Eiermann W, Pienkowski T, Martin M, Robert N, Crown J, Nuciforo P, Bee V, Mackey J, Slamon DJ, Press MF. PTEN Loss Is Associated with Worse Outcome in HER2-Amplified Breast Cancer Patients but Is Not Associated with Trastuzumab Resistance. Clin Cancer Res. 2015 May 1;21(9):2065-74. doi: 10.1158/1078-0432.CCR-14-2993. Epub 2015 Feb 3. PMID 25649019
- [Derived] Blasco A, Lopez-Tarruella S, Urruticoechea A, Carrasco E, Spera G, Martin M, Bermejo B, Chap L, Ruiz-Borrego M, Crown J, Garcia-Saenz JA, Chan A, Guerrero-Zotano A, Semiglazov V, Calvo L, Pienkowski T, Herranz J, Slamon D. Intermediate endpoints as surrogates for long-term outcomes in breast cancer adjuvant chemotherapy trials. Oncologist. 2025 Sep 1;30(9):oyaf263. doi: 10.1093/oncolo/oyaf263. PMID 40838872
- [Derived] Press MF, Sauter G, Buyse M, Fourmanoir H, Quinaux E, Tsao-Wei DD, Eiermann W, Robert N, Pienkowski T, Crown J, Martin M, Valero V, Mackey JR, Bee V, Ma Y, Villalobos I, Campeau A, Mirlacher M, Lindsay MA, Slamon DJ. HER2 Gene Amplification Testing by Fluorescent In Situ Hybridization (FISH): Comparison of the ASCO-College of American Pathologists Guidelines With FISH Scores Used for Enrollment in Breast Cancer International Research Group Clinical Trials. J Clin Oncol. 2016 Oct 10;34(29):3518-3528. doi: 10.1200/JCO.2016.66.6693. PMID 27573653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 433 centers in 43 countries. A total of 3222 participants randomized between 05 April 2001 and 30 March 2004. Participants stratified according to institution, nodal status(negative, positive 1-3 nodes, positive 4 or more nodes) and hormonal receptor status (estrogen and/or progesterone receptor positive versus negative).
Pre-assignment Details: Participants were randomized in 1:1:1 ratio to receive adjuvant therapy with either AC→ T, AC→ TH or TCH. During the course of the study, some participants received treatment different from the arm in which they were randomized. The safety analyses was conducted as per the treatment received.
Period: Overall Study
Arm/Group | Doxorubicin+Cyclophosphamide (AC) Followed by Docetaxel (AC→T) | AC Followed by Docetaxel + Herceptin (AC→TH) | Docetaxel + Carboplatin + Herceptin (TCH)
Started | 1073 (Randomized) | 1074 (Randomized) | 1075 (Randomized)
Treated | 1045 | 1072 | 1057
Safety Population | 1018 (1018 participants received AC-T (1012 from AC-T arm, 6 from AC-TH arm).) | 1100 (1100 participants received AC-TH (1066 from AC-TH arm, 33 from AC-T arm and 1 from TCH arm).) | 1056 (1056 participants received TCH.)
Completed | 952 | 804 | 926
Not Completed | 121 | 270 | 149
Not completed — Death | 1 | 0 | 2
Not completed — Breast cancer relapse | 5 | 18 | 11
Not completed — Second primary malignancy | 0 | 4 | 1
Not completed — Withdrawal by Subject | 41 | 64 | 26
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Cardiac toxicity | 0 | 61 | 32
Not completed — Herceptin toxicity | 0 | 22 | 6
Not completed — Adverse Event | 46 | 30 | 18
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Other than specified above | 0 | 38 | 19
Not completed — Missing | 0 | 27 | 13
Not completed — Randomized but not treated | 28 | 2 | 18

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) population included all randomized participants.
Groups:
- Doxorubicin+Cyclophosphamide (AC) Followed by Docetaxel (AC→T): Doxorubicin 60 mg/m² IV bolus injection in combination with cyclophosphamide 600 mg/m² IV bolus injection on Day 1 of every 3 weeks for 4 cycles followed by docetaxel 100 mg/m² IV infusion every 3 weeks for another 4 cycles.
- Total: Total of all reporting groups
Arm/Group | Doxorubicin+Cyclophosphamide (AC) Followed by Docetaxel (AC→T) | AC Followed by Docetaxel + Herceptin (AC→TH) | Docetaxel + Carboplatin + Herceptin (TCH) | Total
Number analyzed (Participants) | 1073 | 1074 | 1075 | 3222
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (9.7) | 48.7 (9.7) | 48.6 (9.9) | 48.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1073 | 1074 | 1075 | 3222
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Free Survival at 5 Years
Description: Disease Free Survival was defined as the interval from the date of randomization to the date of local, regional or metastatic relapse or the date of second primary cancer (with the exception of curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix) or death from any cause whichever occured first. Disease free survival was estimated using the Kaplan-Meier method.
Time Frame: From randomization until relapse or death or up to 5 years
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxorubicin+Cyclophosphamide (AC) Followed by Docetaxel (AC→T) | AC Followed by Docetaxel + Herceptin (AC→TH) | Docetaxel + Carboplatin + Herceptin (TCH)
Number analyzed (Participants) | 1073 | 1074 | 1075
percentage of participants | 75.5 [72.8 to 78.2] | 83.2 [80.9 to 85.4] | 81.0 [78.6 to 83.4]

2. Secondary Outcome: Percentage of Participants With Disease Free Survival at 10 Years
Description: as for outcome 1
Time Frame: From randomization until relapse or death or up to 10 years
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Doxorubicin+Cyclophosphamide (AC) Followed by Docetaxel (AC→T) | AC Followed by Docetaxel + Herceptin (AC→TH) | Docetaxel + Carboplatin + Herceptin (TCH)
Number analyzed (Participants) | 1073 | 1074 | 1075
percentage of participants | 67.2 [64.2 to 70.2] | 73.4 [70.6 to 76.2] | 72.3 [69.4 to 75.1]

3. Secondary Outcome: Overall Survival- Percentage of Participants Who Survived at 10 Years
Description: Overall survival of the participants was measured from the date of randomization up to the date of death due to any cause. Overall survival was estimated using the Kaplan-Meier method.
Time Frame: From randomization until death or up to 10 years
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Doxorubicin+Cyclophosphamide (AC) Followed by Docetaxel (AC→T) | AC Followed by Docetaxel + Herceptin (AC→TH) | Docetaxel + Carboplatin + Herceptin (TCH)
Number analyzed (Participants) | 1073 | 1074 | 1075
percentage of particpants | 78.9 [76.2 to 81.5] | 86.0 [83.8 to 88.2] | 83.4 [81.0 to 85.8]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from the time the participant started treatment with study drug until 30 days after the last infusion of study treatment (chemotherapy or Herceptin).
Description: Reported AEs are treatment-emergent AEs that is AEs that developed/worsened during the 'on treatment period' (from the first infusion of study drug until 30 days after the last infusion of study drug). Safety population included all treated participants. Source vocabulary used to define AE term: Pooled NCI-CTC version 2.0 and COSTART version 5.0
Arm/Group | Doxorubicin+Cyclophosphamide (AC) Followed by Docetaxel (AC→T) | AC Followed by Docetaxel + Herceptin (AC→TH) | Docetaxel + Carboplatin + Herceptin (TCH)
Serious Adverse Events (participants affected / at risk) | 218/1018 | 298/1100 | 283/1056
Other Adverse Events (participants affected / at risk) | 1017/1018 | 1100/1100 | 1052/1056
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin+Cyclophosphamide (AC) Followed by Docetaxel (AC→T) (N=1018) | AC Followed by Docetaxel + Herceptin (AC→TH) (N=1100) | Docetaxel + Carboplatin + Herceptin (TCH) (N=1056)
ANEMIA (Blood and lymphatic system disorders) | 1 | 8 | 9
LEUKOPENIA (Blood and lymphatic system disorders) | 21 | 23 | 20
LYMPHEDEMA (Blood and lymphatic system disorders) | 0 | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 1 | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 3
ANGINA PECTORIS (Cardiac disorders) | 0 | 1 | 1
AORTIC STENOSIS (Cardiac disorders) | 0 | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 2 | 3 | 3
ARTERIAL ANOMALY (Cardiac disorders) | 0 | 0 | 1
AV BLOCK (Cardiac disorders) | 0 | 0 | 1
CARDIOMYOPATHY (Cardiac disorders) | 0 | 2 | 1
CARDIOVASCULAR DISORDER (Cardiac disorders) | 2 | 0 | 0
CAROTID OCCLUSION (Cardiac disorders) | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (Cardiac disorders) | 0 | 1 | 3
DEEP THROMBOPHLEBITIS (Cardiac disorders) | 6 | 13 | 15
ELECTROCARDIOGRAM ABNORMAL (Cardiac disorders) | 0 | 0 | 1
HEART ARREST (Cardiac disorders) | 0 | 2 | 1
HEART FAILURE (Cardiac disorders) | 0 | 1 | 0
HEMORRHAGE (Cardiac disorders) | 0 | 2 | 2
HYPERTENSION (Cardiac disorders) | 0 | 0 | 1
HYPOTENSION (Cardiac disorders) | 0 | 1 | 0
LEFT HEART FAILURE (Cardiac disorders) | 8 | 25 | 2
MYOCARDIAL ISCHEMIA (Cardiac disorders) | 0 | 5 | 4
MYOCARDITIS (Cardiac disorders) | 1 | 0 | 0
PALPITATION (Cardiac disorders) | 0 | 3 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0
PHLEBITIS (Cardiac disorders) | 0 | 1 | 0
POSTURAL HYPOTENSION (Cardiac disorders) | 0 | 1 | 0
SYNCOPE (Cardiac disorders) | 1 | 4 | 1
TACHYCARDIA (Cardiac disorders) | 2 | 0 | 2
VASCULITIS (Cardiac disorders) | 0 | 1 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 1 | 0
THYROID DISORDER (Endocrine disorders) | 1 | 0 | 0
ANOREXIA (Gastrointestinal disorders) | 0 | 0 | 1
CHOLECYSTITIS (Gastrointestinal disorders) | 2 | 0 | 1
CHOLELITHIASIS (Gastrointestinal disorders) | 0 | 2 | 1
COLITIS (Gastrointestinal disorders) | 0 | 1 | 4
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 1
DIARRHEA (Gastrointestinal disorders) | 2 | 10 | 11
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1
ESOPHAGITIS (Gastrointestinal disorders) | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 1 | 0
GASTROENTERITIS (Gastrointestinal disorders) | 1 | 2 | 3
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
HEMATEMESIS (Gastrointestinal disorders) | 0 | 1 | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 0 | 1
MELENA (Gastrointestinal disorders) | 1 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 7 | 3
PERFORATED STOMACH ULCER (Gastrointestinal disorders) | 0 | 1 | 0
PROCTITIS (Gastrointestinal disorders) | 0 | 0 | 1
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
STOMACH ULCER (Gastrointestinal disorders) | 0 | 0 | 2
STOMATITIS (Gastrointestinal disorders) | 7 | 4 | 1
VOMITING (Gastrointestinal disorders) | 12 | 16 | 11
ABDOMINAL PAIN (General disorders) | 2 | 3 | 2
ABSCESS (General disorders) | 0 | 0 | 1
ACCIDENTAL INJURY (General disorders) | 0 | 3 | 3
AGGRAVATION REACTION (General disorders) | 0 | 0 | 1
ALLERGIC REACTION (General disorders) | 2 | 7 | 5
ASTHENIA (General disorders) | 4 | 3 | 6
BACK PAIN (General disorders) | 1 | 3 | 0
CELLULITIS (General disorders) | 7 | 7 | 11
CHEST PAIN (General disorders) | 5 | 7 | 6
CHILLS (General disorders) | 1 | 0 | 0
CYST (General disorders) | 0 | 0 | 4
FEVER (General disorders) | 85 | 109 | 86
HEADACHE (General disorders) | 1 | 0 | 1
HYPOTHERMIA (General disorders) | 0 | 1 | 0
IMMUNE SYSTEM DISORDER (General disorders) | 0 | 1 | 0
INFECTION (General disorders) | 68 | 85 | 85
INJECTION SITE PAIN (General disorders) | 0 | 0 | 1
MUCOUS MEMBRANE DISORDER (General disorders) | 0 | 0 | 1
PAIN (General disorders) | 1 | 1 | 0
PERITONITIS (General disorders) | 0 | 0 | 1
PHOTOSENSITIVITY REACTION (General disorders) | 0 | 1 | 0
RADIATION INJURY (General disorders) | 0 | 1 | 0
REACTION UNEVALUABLE (General disorders) | 0 | 0 | 1
SEPSIS (General disorders) | 0 | 0 | 1
DEAFNESS (General disorders) | 0 | 1 | 0
EAR PAIN (General disorders) | 1 | 0 | 0
OTITIS MEDIA (General disorders) | 0 | 1 | 0
VESTIBULAR DISORDER (General disorders) | 0 | 1 | 0
ACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 5 | 5
EDEMA (Metabolism and nutrition disorders) | 0 | 0 | 1
ENZYMATIC ABNORMALITY (Metabolism and nutrition disorders) | 0 | 1 | 0
GENERALIZED EDEMA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 | 0 | 2
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 0 | 0 | 3
HYPONATREMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOVOLEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
PERIPHERAL EDEMA (Metabolism and nutrition disorders) | 1 | 1 | 1
SGOT INCREASED (Metabolism and nutrition disorders) | 0 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
JOINT DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
ANXIETY (Nervous system disorders) | 1 | 1 | 0
CEREBRAL INFARCT (Nervous system disorders) | 0 | 1 | 0
COMA (Nervous system disorders) | 0 | 0 | 1
CONFUSION (Nervous system disorders) | 0 | 1 | 0
CONVULSION (Nervous system disorders) | 0 | 0 | 1
DEPRESSION (Nervous system disorders) | 0 | 5 | 3
DIZZINESS (Nervous system disorders) | 0 | 1 | 0
EMOTIONAL LABILITY (Nervous system disorders) | 0 | 2 | 0
GRAND MAL CONVULSION (Nervous system disorders) | 0 | 1 | 0
MENINGITIS (Nervous system disorders) | 1 | 0 | 0
NEUROPATHY (Nervous system disorders) | 3 | 3 | 4
TRISMUS (Nervous system disorders) | 0 | 0 | 1
VERTIGO (Nervous system disorders) | 0 | 0 | 2
BREAST NEOPLASM (Renal and urinary disorders) | 0 | 1 | 1
CYSTITIS (Renal and urinary disorders) | 0 | 1 | 0
ENDOMETRIAL CARCINOMA (Renal and urinary disorders) | 0 | 1 | 0
ENDOMETRIAL DISORDER (Renal and urinary disorders) | 1 | 0 | 0
HEMATURIA (Renal and urinary disorders) | 0 | 0 | 2
KIDNEY FAILURE (Renal and urinary disorders) | 0 | 0 | 1
KIDNEY FUNCTION ABNORMAL (Renal and urinary disorders) | 0 | 0 | 1
MENSTRUAL DISORDER (Renal and urinary disorders) | 0 | 0 | 1
TOXIC NEPHROPATHY (Renal and urinary disorders) | 0 | 1 | 0
URINARY TRACT DISORDER (Renal and urinary disorders) | 0 | 0 | 1
URINARY TRACT INFECTION (Renal and urinary disorders) | 0 | 2 | 1
VAGINITIS (Renal and urinary disorders) | 0 | 0 | 1
APNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
LUNG EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
LUNG FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 3
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
ACNE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
APPLICATION SITE REACTION (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
EXFOLIATIVE DERMATITIS (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
FUNGAL DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
MACULOPAPULAR RASH (Skin and subcutaneous tissue disorders) | 4 | 1 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
SKIN BENIGN NEOPLASM (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin+Cyclophosphamide (AC) Followed by Docetaxel (AC→T) (N=1018) | AC Followed by Docetaxel + Herceptin (AC→TH) (N=1100) | Docetaxel + Carboplatin + Herceptin (TCH) (N=1056)
LYMPHEDEMA (Blood and lymphatic system disorders) | 81 | 94 | 107
HYPERTENSION (Cardiac disorders) | 40 | 72 | 78
LEFT HEART FAILURE (Cardiac disorders) | 30 | 71 | 31
PALPITATION (Cardiac disorders) | 69 | 94 | 95
TACHYCARDIA (Cardiac disorders) | 50 | 62 | 67
ANOREXIA (Gastrointestinal disorders) | 230 | 238 | 252
CONSTIPATION (Gastrointestinal disorders) | 383 | 403 | 351
DIARRHEA (Gastrointestinal disorders) | 439 | 555 | 658
DYSPEPSIA (Gastrointestinal disorders) | 204 | 273 | 263
NAUSEA (Gastrointestinal disorders) | 890 | 967 | 863
STOMATITIS (Gastrointestinal disorders) | 660 | 735 | 564
VOMITING (Gastrointestinal disorders) | 563 | 628 | 428
ABDOMINAL PAIN (General disorders) | 179 | 220 | 240
ALLERGIC REACTION (General disorders) | 100 | 137 | 153
ASTHENIA (General disorders) | 838 | 925 | 878
BACK PAIN (General disorders) | 82 | 132 | 96
CHEST PAIN (General disorders) | 73 | 103 | 91
CHILLS (General disorders) | 58 | 88 | 78
FEVER (General disorders) | 162 | 206 | 145
HEADACHE (General disorders) | 301 | 323 | 306
INFECTION (General disorders) | 350 | 445 | 327
INJECTION SITE REACTION (General disorders) | 66 | 70 | 84
PAIN (General disorders) | 222 | 268 | 217
AMBLYOPIA (General disorders) | 34 | 52 | 55
CONJUNCTIVITIS (General disorders) | 111 | 122 | 45
DRY EYES (General disorders) | 41 | 56 | 30
LACRIMATION DISORDER (General disorders) | 210 | 264 | 124
TASTE PERVERSION (General disorders) | 291 | 312 | 320
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 77 | 85 | 79
PERIPHERAL EDEMA (Metabolism and nutrition disorders) | 339 | 405 | 347
WEIGHT GAIN (Metabolism and nutrition disorders) | 197 | 262 | 254
WEIGHT LOSS (Metabolism and nutrition disorders) | 81 | 100 | 69
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 439 | 515 | 335
BONE PAIN (Musculoskeletal and connective tissue disorders) | 187 | 235 | 144
MYALGIA (Musculoskeletal and connective tissue disorders) | 541 | 614 | 415
ANXIETY (Nervous system disorders) | 86 | 78 | 70
DEPRESSION (Nervous system disorders) | 106 | 139 | 119
DIZZINESS (Nervous system disorders) | 112 | 154 | 130
DRY MOUTH (Nervous system disorders) | 87 | 55 | 37
EMOTIONAL LABILITY (Nervous system disorders) | 56 | 65 | 41
INSOMNIA (Nervous system disorders) | 226 | 288 | 252
NEUROPATHY (Nervous system disorders) | 514 | 569 | 406
VASODILATATION (Nervous system disorders) | 364 | 416 | 384
BREAST PAIN (Renal and urinary disorders) | 53 | 59 | 62
DYSURIA (Renal and urinary disorders) | 24 | 51 | 58
MENSTRUAL DISORDER (Renal and urinary disorders) | 368 | 356 | 384
COUGH INCREASED (Respiratory, thoracic and mediastinal disorders) | 187 | 205 | 147
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 227 | 270 | 229
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 60 | 143 | 170
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 74 | 94 | 60
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 175 | 277 | 193
ALOPECIA (Skin and subcutaneous tissue disorders) | 1003 | 1083 | 1018
DRY SKIN (Skin and subcutaneous tissue disorders) | 76 | 101 | 61
EXFOLIATIVE DERMATITIS (Skin and subcutaneous tissue disorders) | 87 | 87 | 32
MACULOPAPULAR RASH (Skin and subcutaneous tissue disorders) | 275 | 354 | 330
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 507 | 484 | 303
PRURITUS (Skin and subcutaneous tissue disorders) | 38 | 50 | 66
RASH (Skin and subcutaneous tissue disorders) | 238 | 279 | 313
SKIN DISCOLORATION (Skin and subcutaneous tissue disorders) | 65 | 67 | 50
SWEATING (Skin and subcutaneous tissue disorders) | 67 | 67 | 73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.